CLINICAL TRIAL: NCT00891423
Title: A Randomised Controlled Crossover Pilot Study of Meropenem Standard 30 Minute Infusion Versus Prolonged 3 Hour Infusion in Intensive Care Patients
Brief Title: A Study of Meropenem Standard 30 Minute Infusion Versus Prolonged 3 Hour Infusion in Intensive Care Unit (ICU) Patients
Acronym: MERO001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Health (Other Government)
Responsible Party: Principal Investigator, Katherine Langan, Infectious diseases registrar, Austin Health
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H2008/03406; ACTRN (Registry Identifier: 12612000284864)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Sepsis
Keywords: Meropenem; extended infusion; prolonged infusion; Time above MIC
MeSH Terms: conditions — Sepsis | interventions — Meropenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meropenem short infusion (Active Comparator): Meropenem 1g infused over 30 minutes
  * every 8 hours if calculated CrCL greater than or equal to 50 mL/min OR
  * every 12 hours if calculated CrCL less than 50 mL/min or hemofiltration
  Interventions: Drug: Meropenem short infusion
- Meropenem extended infusion (Experimental): Meropenem 500mg infused over 3 hours
  * every 8 hours if calculated CrCL greater than or equal to 50 mL/min OR
  * every 12 hours if calculated CrCL less than 50 mL/min or hemofiltration
  Interventions: Drug: Meropenem extended infusion

INTERVENTIONS:
Drug: Meropenem short infusion
  Other Names: Merrem
  Arms: Meropenem short infusion
Drug: Meropenem extended infusion
  Other Names: Merrem
  Arms: Meropenem extended infusion

SUMMARY:
Meropenem is a powerful antibiotic used in intensive care for people who have very serious infections. Meropenem is rapidly removed from the blood by the kidneys and it is very expensive. In very ill patients in intensive care, it is uncertain how best to give this antibiotic. Studies have suggested that a smaller dose given over a longer period of time, results in blood levels of meropenem that are just as good as when a higher dose is given over a shorter period of time. This direct comparison has not been tested in intensive care patients. It is important to know this because if giving a lesser amount more slowly is just as good, then doctors will choose to give meropenem this way. To establish whether this is the case, the investigators plan to conduct an initial (pilot) study in ten intensive care patients at Austin hospital.

Adult (age 18 years or older) patients in intensive care who have a serious infection being treated with the antibiotic, meropenem for three days or more will be able to participate in this study. The decision to start meropenem will be made by the intensive care doctors and they will give it in the usual way for 24 hours.

The investigators will then in a random way (like tossing of a coin), give the participant meropenem either in the usual way (1 gram infused over 30 minutes) or give them a smaller amount, but over a longer period of time (500 milligrams infused over 3 hours). This will be done for 24 hours. They will then receive meropenem in the alternative way for another 24 hours. After this time the intensive care doctors will decide how meropenem will continue to be given.

Blood levels of meropenem will be measured to see if they are the same when meropenem is given in each of the two different ways. During each different way of giving meropenem, 7 blood samples will need to be taken. Ten mls (or one spoonful) of blood will be required for each measurement. Blood levels will be taken through monitoring lines, which will be already present.

Other information will also be collected about the participant during this study. This will include their age, gender, height, weight, information about what other medical conditions they have and measurements of how well their kidneys are functioning.

DETAILED DESCRIPTION:
The use of pharmacodynamic and pharmacokinetic principles in antibiotic dosing is advocated to enable more effective and efficient use of antibiotics.

The current standard of care in Austin ICU is to give meropenem 1g via short (30 min) infusion. Small studies of healthy volunteers and intensive care patients and Monte Carlo simulation modelling in these groups, have shown that prolonged infusions of meropenem can provide at least equivalent T > MIC while using a smaller dose. Studies in intensive care patients have generally excluded those with renal failure, septic shock and certain other co-morbidities. Therefore, a study encompassing all groups of patients who receive meropenem in the intensive care setting is required to show if these findings have more generalised applicability.

Hypothesis/research questions:

500mg of meropenem administered as a 3 hour infusion is at least comparable to more traditional dosing of 1 g administered as a 30 minute infusion, in attaining target time above MIC.

We plan to compare standard meropenem therapy (1g over 30 minute infusion) with prolonged infusion meropenem (500mg over 3 hour infusion) in a general intensive care unit. Meropenem levels will be monitored by high performance liquid chromatography (HPLC) analysis (Victorian College of Pharmacy) to determine pharmacokinetic and pharmacodynamic outcomes of the different dosing regimens and will be correlated with the meropenem MIC of any significant bacterial isolates from the patients

The outcomes of this pilot study will help plan a larger project to improve the use of meropenem in intensive care unit patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult intensive care patients
* Predicted duration of treatment 3 days or more

Exclusion Criteria:

* Predicted duration of treatment less than 3 days
* Hypersensitivity to meropenem or other beta-lactams
* Consent unable to be obtained by participant or next of kin
* Suspected or proven bacterial meningitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-04; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Time above MIC | 01/31/2010

CONTACTS AND LOCATIONS:
Overall Officials: Paul JOHNSON, Study Director — Austin Health
Locations (1):
- Austin Health, Melbourne, Victoria, Australia